CLINICAL TRIAL: NCT05381259
Title: Effectiveness of Hortitherapy on the Immediate Well-being of Elderly People With Alzheimer's Disease or Related in Day Care
Acronym: Hortitherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Médical Porte Verte (Other)
Responsible Party: Principal Investigator, Adèle de Malherbe, Study coordinator, Centre Médical Porte Verte
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-A00357-36
Record Dates: First submitted 2022-05-03; First posted 2022-05-19 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-05

CONDITIONS: Horticultural Therapy

STUDY DESIGN:
Intervention Model Description: Part of the group having agreed to participate in the study will carry out the horticultural workshop while the other group will benefit from the workshop usually offered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hortitherapy intervention versus control (Other): Horticultural therapy refers to physical and psychic therapy by nature by focusing on the action of gardening on the body, intellect, psych and mind.
  Horticultural in the form of therapeutic gardening serves as a support to help and treat various pathologies in the brain.
  It is a form of curative treatment exploiting the planting and maintenance of garden. The term is a contraction of " horticultural " and " therapy".
  Interventions: Behavioral: hortitherapy in people living with Alzheimer's taking place in three different day care

INTERVENTIONS:
Behavioral: hortitherapy in people living with Alzheimer's taking place in three different day care — 6 users benefiting from the horticultural workshop and 6 others from a usual workshop (control group) This control group will benefit from its usual workshop while the other group will participate in the horticultural workshop.
  If it is impossible to carry out the workshops outdoors (rain or high heat), the day reception centers will provide a room to allow the workshops to be carried out. They will be adapted in terms of activities and materials.

SUMMARY:
Currently, there are an estimated 47 million people with dementia worldwide, with approximately 10 million new cases diagnosed each year. This figure is expected to triple to 130 million in 2050.

In France, the number of dementia cases is estimated at 754,000 and could reach 1,813,000 in 2050.

In a recent literature review, researchers highlighted the many benefits of horticultural therapy and garden environments for people with Alzheimer's or cognitive disorders. They include: alleviating pain, improving attention, decreasing stress, relieving agitation, decreasing the use of medications, such as antipsychotics, as well as reducing falls.

Gardening offers a non-pharmacological approach to achieving these goals and could improve the quality of life for people with Alzheimer's disease or another dementia. As part of a care solution, support services that include social activities, such as gardening, reduce the need for more intrusive and expensive care solutions.

The objective of this research is to evaluate the impact of horticultural

DETAILED DESCRIPTION:
This research is an interventional study involving the human person of category 2 involving only minimal risks and constraints, it is prospective, multicenter and non-randomized.

The study will take place with users of the Lépine Versailles day care centre, the La Porte Verte hospital and the Les Magnolias Geriatric Center, living with cognitive disorders. For the purposes of this study, understanding the instructions is required.

The people welcomed will participate in their usual day supervised by the day reception team.

Part of the group having agreed to participate in the study will carry out the horticultural workshop while the other group will benefit from the workshop usually offered. The study will be done with 52 users with the participation of a supervisor to animate the workshops of the different groups.

Each site will have a workshop that will take place in the morning from 11 a.m. to 12 p.m. and one in the afternoon from 2:30 p.m. to 3:30 p.m. This will make it possible to compare the well-being of users according to the time of the workshop.

ELIGIBILITY:
Inclusion Criteria:

* Patient having signed an informed and written consent,
* Patient aged over 60,
* Patient with Alzheimer's or related disease,
* Patient benefiting from day care,
* Patient under guardianship or curatorship.

Exclusion Criteria:

* Patient in period of adaptation in day care,
* Patient in temporary care at day care,
* Patient having participated in less than 4 horticultural workshops during the cycle,
* Patient with severe asthma and/or an allergy that does not allow workshops to be carried out,
* Patient with major behavioral problems that make it impossible to carry out the workshops.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-05-04 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
EVIBE : An instant assessment scale of perceived well-being in people with major cognitive problems. | Eight months
  The score of the EVIBE scale is a numerical score between 0 and 5, it will be compared between the two groups, the patients will be integrated randomly in order to take into account the correlation between the data due to the repeated nature of the measurements.
  The regression application conditions will be checked graphically on the residuals. If they are not respected, alternative strategies will be studied (log transformation, bootstrap test)

SECONDARY OUTCOMES:
Tinetti test : Assessment of walking and balance (Tinetti 1986). | Eight months
  The Tinetti test is an effective and reproducible tool for the assessment of the risk of falling, its administration time is approximately 5 to 10 minutes and evaluates static and dynamic balance.
HAD Scale : Hospital Anxiety and Depression | Eight months
  The advantage of this scale is to quickly and simultaneously assess depressive and anxious dimensions using a short questionnaire. The scale is collected on inclusion and after the 8 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Adèle DE MALHERBE, Dr, Study Director — Director of the Medico-Social Departement; Benjamin BAUBERT, Principal Investigator — CENTRE 2 EHPAD Lépine Versailles; ophelie LEMBRET, Principal Investigator — CENTRE 3 HPGM
Locations (1):
- CentreMédicalPorteVerte, Versailles, France